CLINICAL TRIAL: NCT02354092
Title: Paracervical Block for Pain Control During Osmotic Dilator Placement: a Randomized Controlled Trial
Brief Title: Paracervical Block for Pain Control With Osmotic Dilator Placement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Principal Investigator, Lisa Bayer, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141593
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Abortion Late; Pain
Keywords: cervical dilation; pain; paracervical block; osmotic dilators
MeSH Terms: conditions — Pain | interventions — Anesthetics, Local; salicylhydroxamic acid; Anesthesia, Obstetrical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Group (Sham Comparator): This non-intervention group will receive the sham paracervical block. This intervention will include
  * Preprocedural pain control: 800 mg Ibuprofen prior to dilator placement
  * Local anesthetic for tenaculum placement
  * Sham Paracervical Block done with capped spinal needle
  * osmotic dilators placed in the usual fashion
  * postprocedural assessment
  Interventions: Procedure: Local anesthetic for tenaculum placement; Procedure: Sham; Procedure: Dilator Placement; Behavioral: Post-procedural assessment; Drug: Preprocedural pain control
- Paracervical Block Group (Experimental): This intervention group will receive the paracervical block. This intervention will include
  * Preprocedural pain control: 800 mg Ibuprofen prior to dilator placement
  * Local anesthetic for tenaculum placement
  * 18 ml 1% buffered lidocaine Paracervical Block
  * osmotic dilators placed in the usual fashion
  * postprocedural assessment
  Interventions: Procedure: Local anesthetic for tenaculum placement; Procedure: Paracervical Block; Procedure: Dilator Placement; Behavioral: Post-procedural assessment; Drug: Preprocedural pain control

INTERVENTIONS:
Procedure: Local anesthetic for tenaculum placement — 2 mL of buffered Lidocaine injected superficially at anterior lip of cervix in 12 o'clock position Drug: 1% Lidocaine Hydrochloride, 8.4% Sodium Bicarbonate
Procedure: Sham — Over 60 seconds, without moving the tenaculum, a capped needle gently touches the vaginal sidewall at the level of the external os at 4 and 8 o'clock positions
  Arms: Sham Group
Procedure: Paracervical Block — 18 mL of buffered Lidocaine is slowly injected into the vaginal fornices and equally distributed at 4 and 8 o'clock. The injection is continuous from superficial to deep (3cm) to superficial (injecting with insertion and withdrawal) Drug: 1% Lidocaine Hydrochloride, 8.4% Sodium Bicarbonate
  Arms: Paracervical Block Group
Procedure: Dilator Placement — Osmotic dilators will be placed in the usual fashion with a combination of Dilapan-S and laminaria per clinician preference
  Drugs:
  Dilapan-S is a hygroscopic cervical dilator made of a patented hydrogel called AQUACRYL. It is a rigid hydrophilic stick that increases in volume by absorbing fluids and comfortably dilating the cervix.
  Laminaria is an herbal medicine used to induce labor and abortion. The dried stem of Laminaria mechanically dilates the cervical opening by absorbing water and swelling to several times its original diameter.
Behavioral: Post-procedural assessment — 15 minutes after procedure, subjects will complete a questionnaire that collects information about pain, negative symptoms, and assessment of how effective their pain management was.
Drug: Preprocedural pain control — 800 mg Ibuprofen taken before dilator placement

SUMMARY:
Cervical dilators are frequently used for preparation prior to second trimester surgical abortion. While their use decreases complications associated with surgical abortion, their placement is often uncomfortable for the patient. Currently there are no proven methods for reducing pain during osmotic dilator placement. The use of numbing medication around the cervix (paracervical block) may decrease this placement pain.

DETAILED DESCRIPTION:
It is estimated that 1.21 million abortions were performed in 2008. Of these, approximately 11% occurred in the second trimester and 1.4% occurred after 21 weeks gestation. In the United States, dilation and evacuation (D&E) is the most common method of terminating a second trimester pregnancy with greater than 98% of second trimester abortions occurring by D&E.

Pre-procedure cervical preparation decreases the incidence of complications associated with D&E. Cervical dilators are often used prior to second trimester D&Es to aid in softening and dilating the cervix. Typically, dilator placement occurs the day of the D&E or 1-2 days prior and oftentimes occurs in an outpatient clinic setting without anesthesia readily available. Many women experience moderate to severe discomfort with osmotic dilator insertion. Providers use various methods to minimize this discomfort including paracervical block (PCB), non-steroidal anti-inflammatory medications (NSAIDs), anxiolytics and narcotics. In particular, PCB and NSAIDs are readily available in the clinic setting and can be used for this purpose. There is, however, no data to support their efficacy in ameliorating the pain of dilator insertion.

Paracervical blocks are used commonly to decrease pain in abortion procedures and other gynecological procedures. The PCB is thought to work primarily by blocking pain conduction via Frankenhauser's plexus. As such, their effect may be most important in relieving the pain associated with cervical dilation. In a recent randomized control trial, PCB prior to first trimester surgical abortion was found to significantly reduce pain with cervical dilation and uterine aspiration. Since osmotic dilator placement primarily involves cervical manipulation and dilation, PCB may provide some pain relief over placebo. The research team proposes a randomized controlled trial to evaluate the efficacy of a PCB in decreasing pain associated with osmotic dilator placement. This trial will also provide information about the degree of pain that women experience during osmotic dilator placement; information not previously known.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily seeking surgical pregnancy termination
* gestational age on day of study 14w0d to 23w6d confirmed by pelvic ultrasound with a viable pregnancy (no fetal demise diagnosed)
* eligible for second trimester D&E
* having osmotic dilators placed for cervical preparation the day prior to D&E
* able and willing to give informed consent and agree to terms of the study
* able to speak and read English or Spanish

Exclusion Criteria:

* took any prescription or illegal drugs 24 hours prior to the appointment
* drank alcohol 12 hours prior to the appointment
* took any over the counter pain medications 12 hours prior to the appointment other than the standard 800mg of Ibuprofen
* contraindications to osmotic dilators
* allergic reaction or hypersensitivity to NSAIDs or lidocaine
* untreated acute cervicitis or pelvic inflammatory disease
* weight <100 pounds

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2015-08-25 (Actual); Study Completion 2015-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bayer, MD MPH, Principal Investigator — UCSD Department of Reproductive Medicine; Sheila Mody, MD MPH, Principal Investigator — UCSD Department of Reproductive Medicine; Kelly Culwell, MD MPH, Principal Investigator — Planned Parenthood of the Pacific Southwest
Locations (2):
- United States (2):
  - Planned Parenthood of the Pacific Southwest: First Avenue Family Planning Michelle Wagner Center, San Diego, California
  - UCSD Medical Offices South: Women's Health Services, San Diego, California

REFERENCES:
- [Background] Glantz JC, Shomento S. Comparison of paracervical block techniques during first trimester pregnancy termination. Int J Gynaecol Obstet. 2001 Feb;72(2):171-8. doi: 10.1016/s0020-7292(00)00292-7. PMID 11166751
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Jones RK, Zolna MR, Henshaw SK, Finer LB. Abortion in the United States: incidence and access to services, 2005. Perspect Sex Reprod Health. 2008 Mar;40(1):6-16. doi: 10.1363/4000608. PMID 18318867
- [Background] Peterson WF, Berry FN, Grace MR, Gulbranson CL. Second-trimester abortion by dilatation and evacuation: an analysis of 11,747 cases. Obstet Gynecol. 1983 Aug;62(2):185-90. PMID 6866362
- [Background] Cansino C, Edelman A, Burke A, Jamshidi R. Paracervical block with combined ketorolac and lidocaine in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2009 Dec;114(6):1220-1226. doi: 10.1097/AOG.0b013e3181c1a55b. PMID 19935022
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Schulz KF, Grimes DA, Cates W Jr. Measures to prevent cervical injury during suction curettage abortion. Lancet. 1983 May 28;1(8335):1182-5. doi: 10.1016/s0140-6736(83)92464-9. PMID 6133988
- [Background] Strauss LT, Gamble SB, Parker WY, Cook DA, Zane SB, Hamdan S; Centers for Disease Control and Prevention. Abortion surveillance--United States, 2003. MMWR Surveill Summ. 2006 Nov 24;55(11):1-32. PMID 17119534
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Group | Paracervical Block Group
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Group | Paracervical Block Group | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (4.3) | 27.6 (7.2) | 25.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Pain at Time of Osmotic Dilator Placement
Description: Measure of distance (mm) from the left ("no pain") on the 100-mm visual analog scale (VAS - reflecting magnitude of pain) recorded at time immediately after osmotic dilator placement. 0 mm=No Pain and 100 mm= worst possible pain. A higher score indicates a higher level of pain.
Time Frame: Within 5 minutes of PCB or sham procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Group | Paracervical Block Group
Number analyzed (Participants) | 7 | 7
units on a scale | 46 (37) | 32 (30)

2. Secondary Outcome: Pain With Paracervical Block or Sham
Description: Measure of distance (mm) from the left ("no pain") on the 100-mm visual analog scale (VAS - reflecting magnitude of pain) recorded at time immediately after last injection for paracervical block OR script for sham injection. 0 mm=No Pain and 100 mm= worst possible pain. A higher score indicates a higher level of pain.
Time Frame: Within 5 minutes after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Group | Paracervical Block Group
Number analyzed (Participants) | 7 | 7
units on a scale | 19 (21) | 39 (18)

3. Secondary Outcome: Reported Pain at Baseline
Description: Measure of distance (mm) from the left ("no pain") on the 100-mm visual analog scale (VAS - reflecting magnitude of pain) of pain recorded at baseline prior to the paracervical block or sham block procedure. 0 mm=No Pain and 100 mm= worst possible pain. A higher score indicates a higher level of pain.
Time Frame: Baseline, just prior to PCB or sham procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Group | Paracervical Block Group
Number analyzed (Participants) | 7 | 7
units on a scale | 4 (4) | 19 (29)

4. Secondary Outcome: Pain With Overall Dilator Placement
Description: Measure of distance (mm) from the left ("no pain") on the 100-mm visual analog scale (VAS - reflecting magnitude of pain) recorded 15 minutes after osmotic dilator placement. mm=No Pain and 100 mm= worst possible pain. A higher mean score indicates a higher level of pain experienced at this time point.
Time Frame: 15 minutes after dilator placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Group | Paracervical Block Group
Number analyzed (Participants) | 7 | 7
units on a scale | 42 (30) | 35 (23)

ADVERSE EVENTS:
Arm/Group | Sham Group | Paracervical Block Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No